CLINICAL TRIAL: NCT05290857
Title: Post-Bleed Management of Antithrombotic Therapy After Gastrointestinal Bleeding: Pilot Study and Registry (PANTHER-GI)
Brief Title: Anticoagulation After GI Bleeding Pilot Study and Registry
Acronym: PANTHER-GI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3349 20210798-01H
Record Dates: First submitted 2022-02-06; First posted 2022-03-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: GastroIntestinal Bleeding; Anticoagulant-induced Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, cohort management study and parallel registry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High thrombotic risk (Experimental): For patients at high thrombotic risk, DOACs will be resumed within 7 days of clinical hemostasis after GI bleeding.
  Interventions: Other: Restart DOAC within 7 days of clinical hemostasis after GI bleeding
- Moderate thrombotic risk (Experimental): For patients at moderate thrombotic risk, DOACs will be resumed between 7 and 14 days of clinical hemostasis after GI bleeding.
  Interventions: Other: Restart DOAC between 7 to 14 days of clinical hemostasis after GI bleeding

INTERVENTIONS:
Other: Restart DOAC within 7 days of clinical hemostasis after GI bleeding — In patients at high thrombotic risk, DOACs will be resumed within 7 days of clinical hemostasis (as judged by the clinical team).
  High thrombotic risk includes the following:
  (i) Atrial fibrillation or atrial flutter with CHA2DS2VASc score of 5 or higher (ii) Atrial fibrillation or atrial flutter with CHA2DS2VASc score or 3 to 4 with recent ischemic stroke, TIA or systemic embolism (within 6 months) (iii) VTE (proximal DVT or PE) within 3 months (iv) Recurrent VTE (proximal DVT or PE) (v) VTE (proximal DVT or PE) associated with antiphospholipid syndrome (if eligible for DOAC) (vi) VTE (proximal DVT or PE) associated with active non-GI cancer (vii) None of the above but considered high thrombotic risk as per investigator
  Arms: High thrombotic risk
Other: Restart DOAC between 7 to 14 days of clinical hemostasis after GI bleeding — In patients at moderate thrombotic risk, DOACs will be resumed between 7 and 14 days of clinical hemostasis (as judged by the clinical team).
  Moderate thrombotic risk includes the following:
  (i) Atrial fibrillation or atrial flutter with CHA2DS2VASc score of 3 to 4 (ii) VTE (proximal DVT or PE) beyond 3 months
  The type and dose of DOAC will be according to patient and physician choice and will be prescribed by the clinical care team.
  Arms: Moderate thrombotic risk

SUMMARY:
PANTHER-GI Pilot Study will assess the feasibility of a full-scale multicentre cohort management study evaluating the safety of a standardized strategy for resuming direct oral anticoagulants (DOACs) after major DOAC-related gastrointestinal (GI) bleeding among patients at moderate to high risk of re-bleeding and thrombosis. A parallel registry will assess whether eligible patients who are not enrolled in the PANTHER-GI Pilot Study are systematically different than enrolled patients and to explore barriers to enrolment.

DETAILED DESCRIPTION:
This pilot cohort management study will evaluate a protocolized strategy for resuming DOACs after major GI bleeding based on thrombotic risk among patients at moderate to high risk of rebleeding. The timeframe for resuming DOACs will be determined based on the patient's underlying thrombotic risk.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older
2. Hospitalized with acute major non-variceal GI bleeding (defined as per ISTH criteria) while receiving OAC therapy (warfarin or DOAC).
3. OAC therapy discontinued for current acute GI bleed and not yet resumed
4. Ongoing indication for long-term anticoagulation of atrial fibrillation (moderate to high risk of stroke/systemic embolism with CHA2DS2VASc score of 3 or higher) or VTE (as per clinical care team)
5. Planned to resume DOAC post-bleed
6. At moderate to high risk of re-bleeding as per clinical care team
7. Clinical hemostasis achieved as per clinical care team
8. Able and willing to comply with follow-up examinations contained within the consent form

Exclusion Criteria:

1. Mechanical heart valve
2. VTE in the context of major transient risk factor and completed 3 months of treatment
3. GI bleeding managed surgically (e.g. gastrectomy, colectomy)
4. Active or previously treated gastrointestinal cancer
5. Life expectancy from other causes of less than 3 months
6. Platelet count < 50,000/µL (or < 50x109/L)
7. Renal dysfunction (Creatine Clearance <30 mL/min as calculated by the Cockcroft-Gault formula)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 18 months
  The pilot study will be considered a success and to have demonstrated feasibility if average recruitment of 2 patients per month at each site is achieved.
Total recruitment | 18 months
  Feasibility criterion of achieving recruitment of 85% of the target sample size of 100 patients

SECONDARY OUTCOMES:
eligibility | 18 months
  proportion of patients screened who are eligible to participate out of all patients screened
consent | 18 months
  proportion of eligible patients who provide consent to participate out of all eligible patients
completion of all required study procedures | 18 months
  proportion of patients who complete all required study procedures out of all enrolled patients
adherence | 18 months
  proportion of patients who adhere to study treatment strategy (i.e. resumed DOAC within the specified timeframe) out of the total number of patients enrolled
repeat endoscopy | 90 days
  proportion of patients with repeat endoscopy for suspected bleeding after index GI bleed out of all enrolled patients
re-hospitalization | 90 days
  number of patients re-hospitalization for GI bleeding after index GI bleed out of all patients enrolled
major bleeding | 90 days
  number of patients with major bleeding (as per International Society on Thrombosis and Haemostasis [ISTH] criteria) out of all patients enrolled
clinically relevant non-major bleeding | 90 days
  number of patients with clinically relevant non-major bleeding (CRNMB; as per ISTH) out of all patients enrolled
acute ischemic stroke, transient ischemic attack or systemic embolism | 90 days
  number of patients who experience composite of acute ischemic stroke, transient ischemic attack or systemic embolism our of all patients enrolled
acute symptomatic VTE | 90 days
  number of patients with acute objectively confirmed venous thromboembolism (symptomatic proximal lower extremity deep vein thrombosis [DVT], symptomatic pulmonary embolism [PE] as per ISTH) out of all patients enrolled
net clinical benefit outcome rate | 90 days
  number of patients experiencing composite of stroke, systemic embolic event, major bleeding, or death from any cause out of all patients enrolled
all-cause mortality | 90 days
  number of patients who die of all causes out of all patients enrolled
functional status | 90 days
  Change in functional status measured using Standard Assessment of Global Activities in the Elderly (SAGE) scale at 90 days compared to baseline.
  SAGE is a 15-item scale that represents a measure of activities of daily living (ADL) across the spectrum of functioning (cognitive, instrumental and basic ADL). The SAGE is supplemented with additional measures of cognition, mood, and quality of life.
  The minimum SAGE score - which corresponds to no functional impairments - is 0. The maximum SAGE score - which corresponds to severe global functional impairment - is 45.
Quality of life of Panther GI Research participants | 90 days
  Quality of life measured using EuroQol-5D [EQ-5D®] at 90 days compared to baseline.
  The EQ-5D instrument comprises a descriptive system questionnaire and a visual analogue scale (EQ VAS). The questionnaire provides a descriptive profile of a respondent's health state representing the level of reported problems on each of the five dimensions of health (mobility, self-care, usual activities, pain or discomfort, anxiety/depression) that can be converted into a single index value. Average index values (expressed as mean and standard deviation or median and interquartile range depending on skewness) at 90 days will be compared to baseline.
  The EQ VAS elicits an individual's rating of their own overall current health (0-100 scale where 0 is the worst health you can imagine and 100 is best health you can imagine). Average EQ VAS ratings (expressed as mean and standard deviation or median and interquartile range depending on skewness) at 90 days will be compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Siegal, MD MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - Alberta Health Services - Peter Lougheed Center Endoscopy Unit, Calgary, Alberta
  - Ottawa Hospital Research Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No